CLINICAL TRIAL: NCT06898905
Title: Hyperfractionated Dual Equivalent Fractionated (HyDEF) Bridging Radiation Therapy in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma Undergoing T-Cell Redirection Therapy
Brief Title: Hyperfractionated Dual Equivalent Fractionated Radiation Therapy
Acronym: HyDEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000038092; IRG-21-132-60-IRG (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2025-03-18; First posted 2025-03-27 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: HyDEF; bridging radiation; once vs twice daily radiation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dual Hyperfractionated Radiation Therapy (Experimental): All patients enrolled will receive radiation as a bridge to subsequent planned T Cell Directed therapy. The same tumor will be treated daily, with one area receiving once daily and the other receiving twice daily radiation therapy.
  Interventions: Other: Bridging Radiation Therapy

INTERVENTIONS:
Other: Bridging Radiation Therapy — Study seeks to compare the hypofractionated radiation therapy with hyperfractionated treatment within the same tumor. Each participant will be serving as their own control; half their tumor will receive once daily hypofractionated (QD) bridging radiotherapy, and the other half of their tumor will receive twice daily hyperfractionated (BID) bridging radiotherapy. Either schedule is considered standard of care and this study aims to determine which schedule may prove superior between the two standards.

SUMMARY:
This study evaluates the feasibility and safety of a novel method for comparing the effectiveness of hypofractionated versus hyperfractionated radiation therapy in participants with relapsed/refractory diffuse large B-cell lymphoma (R/R DLBCL) undergoing T-cell redirection therapies (CAR T-cell therapy or bispecific antibodies).

DETAILED DESCRIPTION:
The purpose of this study is to assess the feasibility and safety of a novel method to study the relative effectiveness of hypo- vs. hyperfractionated therapy (i.e., once daily vs. twice daily treatment) in patients with R/R DLBCL undergoing T-cell redirection therapies. This trial will serve as proof-of-concept, feasibility, and safety for a novel dual fractionation trial design, treating the same tumor with two fractionation schedules, paving the way for future radiotherapy trial designs and direct comparison of the efficacy of once vs. twice daily treatment. Correlative studies of immune exhaustion will evaluate the mechanistic underpinnings between radiotherapy and the immune environment. Finally, with the use of RefleXion BGRT, investigators will collect PET imaging data to provide the basis for this emerging method for administering bridging radiation in lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Adult aged 18 years or older.
4. Histologically confirmed diagnosis of R/R DLBCL with tumor size greater than or equal to 5 cm in its greatest dimension with plan for CAR T or BsAb therapy at Yale New Haven Hospital.
5. ECOG performance status 0 to 3.
6. Ability to present for twice daily (M-F) fractionated radiation therapy, without contraindications for radiotherapy as determined by the treating radiation oncologist.
7. Women of childbearing potential must have a negative serum or urine pregnancy test at screening and at time of radiation treatment planning, per standard of care and departmental standard operating procedure. Participants must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed.

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Participants who are pregnant or currently breastfeeding.

   a. Females who have undergone surgical sterilization or who have been postmenopausal for at least 12 months are not considered to be of childbearing potential.
2. Participants with history of prior radiation exposure for research purposes within the past year, such that participation in this study would place them over the FDA limits for annual radiation exposure.
3. Participants who are unable to safely receive FDG PET tracer.
4. Any condition that would, in the investigator's judgment, interfere with full participation in the study and attending required study visits (if outpatient); pose a significant risk to the participant; or interfere with interpretation of study data.
5. Participants who would not be anticipated to derive any clinical benefit from bridging radiotherapy, are unable to participate in twice daily radiotherapy, or have clinical contraindications to radiation therapy per treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility Assessment of Dual Fractionated Radiation Therapy Enrollment and Treatment | Approximately one year
  The feasibility of the clinical trial's intervention will be assessed based on the ability to enroll and treat at least 5 participants with the proposed dual fractionated radiation therapy, where one half of the tumor receives once daily radiation and the other half receives twice daily radiation. This number is estimated to be sufficient to determine the feasibility of treating a single tumor with different radiation schedules.
Safety analysis of the proposed dual fractionated radiation therapy schema | Throughout the study, approximately two years
  Safety will be assessed by analyzing the incidence of severe (grade ≥ 3) acute toxicities. The therapy will be considered safe if fewer than 30% of study participants receiving dual fractionated radiation therapy experience these toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Robinson, MD PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No